CLINICAL TRIAL: NCT03078465
Title: Ticagrelor Versus High-dose Clopidogrel in Patients With High Platelet Reactivity on Clopidogrel After Percutaneous Coronary Intervention: The PL-PLATELET Randomized Trial
Brief Title: Ticagrelor Versus High-dose Clopidogrel in Patients With High Platelet Reactivity on Clopidogrel After PCI
Acronym: PL-PLATELET
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Competitive studies were conducted at the same time, and enrollment was suspended.
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Shaoliang Chen, MD, Vice President, Nanjing First Hospital, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NFH20170307
Record Dates: First submitted 2017-03-07; First posted 2017-03-13 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Ticagrelor; Clopidogrel

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ticagrelor (Experimental): Administration of ticagrelor 180mg/day for 12 months.
  Interventions: Drug: Ticagrelor
- Clopidogrel (Active Comparator): Administration of clopidogrel 150 mg/day for 12 months
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Ticagrelor — Daily administration of ticagrelor 180mg for 12 months
  Other Names: BRILINTA
  Arms: Ticagrelor
Drug: Clopidogrel — Daily administration of clopidogrel 150mg for 12 months
  Other Names: Plavix, Talcom
  Arms: Clopidogrel

SUMMARY:
To determine the safety and efficacy of Ticagrelor versus Clopidogrel for the reduction of adverse cardiovascular outcomes in patients with high platelet reactivity on clopidogrel after successful implantation of coronary drug-eluting stents.

DETAILED DESCRIPTION:
This is a multi-center, randomized, single-blind, investigator-initiated study with a parallel design. Patients with coronary artery disease undergoing percutaneous coronary intervention and presenting high platelet reactivity on clopidogrel as assessed with the PL-11 analyzer (platelet maximum aggregation ratio [MAR%] ≥ 55 %) at 2 hours post-clopidogrel 300mg LD (Day 0), will be randomized after informed consent, in a 1:1 ratio to the following treatment groups:

Group Α: Ticagrelor 180 mg immediate loading (on Day 0) followed by 180mg/day starting from Day 1 until Day 365 (12 months after randomization).

Group Β: Clopidogrel 150mg per day, starting from Day 1 until Day 365 (12 months after randomization).

Platelet reactivity assessment will be performed before randomization (Day 0), and 3-day after randomization (Day 3). Documentation of major adverse cardiac and cerebrovascular events (death, myocardial infarction, stent thrombosis, stroke, revascularization procedure with PCI or CABG) and serious adverse events (bleeding, other adverse events) will be performed until 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients who agreed to the experimental plan which was permitted by IRB;
* Patients planned to take dual antiplatelet therapy for 12 months.

Exclusion Criteria:

* Severe hepatic dysfunction defined as serum transaminase > 3 times normal limit;
* Renal dysfunction defined as eGFR < 30ml/min/1.73m^2;
* Co-morbidity with an estimated life expectancy of < 50 % at 12 months;
* Scheduled surgery in the next 12 months, which resulted protocol changes;
* Known allergy against study drug or device;
* Use of glycoprotein IIb/IIIa inhibitor during the perioperative period;
* Anticoagulation treatment including warfarin.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2021-05-30 (Estimated); Study Completion 2021-05-30 (Estimated)

PRIMARY OUTCOMES:
12-Month Freedom From MACE | 12 months
  Major adverse cardiovascular and cerebrovascular events consist of all-cause death, target vessel myocardial infarction, stroke, stent thrombosis.

SECONDARY OUTCOMES:
12-Month Freedom From Mortality | 12 months
  All-cause death
12-Month Freedom From Cardiac death | 12 months
  Cardiac death
12-Month Freedom From MI | 12 months
  Myocardial infarction
12-Month Freedom From TLR | 12 months
  Target lesion revascularisation
12-Month Freedom From TVR | 12 months
  Target vessel revascularisation
12-Month Freedom From Stent Thrombosis | 12 months
  Stent thrombus was classified as definite, probable, or possible, according to the definitions provided by the Academic Research Consortium (ARC).Regarding timing, ST was defined as early (<30 days), late (30 days to 1 year), or too late (>1 year).
12-Month Freedom From Stroke | 12 months
  Stroke

OTHER OUTCOMES:
12-Month Freedom From BARC type 2 or above bleeding | 12 months
  BARC (Bleeding Academic Research Consortium) type 2 or above bleeding event following the first dose of study medication
12-Month Freedom From Major or minor bleeding | 12 months
  Major or minor bleeding defined by TIMI (thrombolysis in myocardial infarction) bleeding criteria

CONTACTS AND LOCATIONS:
Overall Officials: Shao-Liang Chen, MD, Study Chair — Nanjing First Hospital, Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang JJ, Gao XF, Ge Z, Tian NL, Liu ZZ, Lin S, Ye F, Chen SL. High platelet reactivity affects the clinical outcomes of patients undergoing percutaneous coronary intervention. BMC Cardiovasc Disord. 2016 Nov 29;16(1):240. doi: 10.1186/s12872-016-0394-0. PMID 27894260